CLINICAL TRIAL: NCT01112774
Title: Investigation of the Mechanisms of Transcranial Direct Current Stimulation of Motor Cortex for the Treatment of Chronic Pain in Spinal Cord Injury
Brief Title: Application of Transcranial Direct Current Stimulation (tDCS) in Patients With Chronic Pain After Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding ended
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010p000190
Record Dates: First submitted 2010-04-20; First posted 2010-04-28 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injury
Keywords: Transcranial direct current stimulation; Spinal cord injury; Chronic pain; Brain excitability
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain | interventions — Transcranial Direct Current Stimulation; Electric Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS/Spinal cord injury (Experimental): Subjects will be randomized to receive 10 sessions of either active or sham tDCS. Stimulation will be given on consecutive days (Monday- Friday) at 2 mA over the primary motor cortex area.
  Interventions: Device: Transcranial direct current stimulation
- tDCS/Healthy subjects (Experimental): Subjects will receive 2 sessions of stimulation: one active and one sham tDCS on two separate visits. The order in which they receive the stimulation will be randomized. Stimulation parameters will be at 2 mA for a total of 20 minutes.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Stimulation will be applied at 2 mA for a total of 20 minutes.
  Other Names: electrical stimulation, tDCS

SUMMARY:
The purpose of this study is to determine whether the novel treatment of transcranial direct current stimulation (tDCS) could decrease the pain perception of those with spinal cord injury.

We will also determine whether these changes are correlated with the clinical outcome (pain reduction).

DETAILED DESCRIPTION:
The active tDCS stimulation sessions will be compared to sham stimulation.

More study details will be provided by Spaulding Rehabilitation Hospital.

ELIGIBILITY:
STUDY ELIGIBILITY CRITERIA (similar to the criteria of the Interstitial Cystitis Network)

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. with traumatic spinal cord injury (complete or incomplete) - for instance, due to fall, car accident or gun shot; (for spinal cord injury only)
4. stable chronic pain for at least the three preceding months(for spinal cord injury only)
5. score higher or equal to 4cm (0 cm= 'no pain' and 10cm='worst possible pain') on the Visual Analogue Scale (VAS) for pain perception at the baseline/start of the treatment(for spinal cord injury only)
6. refractoriness to drugs for pain relieve - such as tricyclic antidepressants, antiepileptic drugs and/or narcotics (pain resistant to at least 2 of these drugs supplied in adequate dosages for six months) (for spinal cord injury only)
7. pain is not attributable to other causes, such as peripheral inflammation.
8. No clinically significant or unstable medical or psychiatric disorder
9. No history of substance abuse
10. No neuropsychiatric comorbidity
11. No implanted devices for pain control, such as vagal or deep brain stimulators
12. No contraindications to tDCS:

    * metal in the head
    * implanted brain medical devices
13. No pregnancy
14. Eligible to MRI according to MRI screening checklist.
15. No use of ventilators

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08-14 (Actual); Study Completion 2013-08-14 (Actual)

PRIMARY OUTCOMES:
Neurophysiological activity changes after treatment with tDCS | baseline, 2 weeks treatment and follow up (2 weeks)
  Magnetic resonance spectroscopy (MRS), electroencephalogram (EEG), transcranial magnetic stimulation (TMS)

SECONDARY OUTCOMES:
Pain changes | Baseline, 2 weeks treatment and follow up (2 weeks)
  (i) Demographic Data; (ii) Visual analog scale (VAS) for pain; (iii) Analgesic use; (iv) Quality of Life Scale (QOLS); (v) Patient Global Assessment (PGA); (vi) Clinical Global Impression (CGI); (vii) Beck Depression Inventory (BDI); (viii) Visual Analog Scale (VAS) for anxiety; (ix) tDCS Side Effects Questionnaire; (x) Mini-mental status exam; and (xi) Validation of Blinding

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States